CLINICAL TRIAL: NCT01576419
Title: Double Blinded, Randomized, Active Drug Comparative, Multi-center, phase3 Clinical Study to Evaluate the Efficacy and Safety of PG201 in Osteoarthritis Patients
Brief Title: Active Drug Comparative, Multi-center, phase3 Clinical Study to Evaluate the Efficacy and Safety of PG201 in Osteoarthritis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PMG Pharm Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PG201-P3
Record Dates: First submitted 2012-04-04; First posted 2012-04-12 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Osteoarthritis of the Knee
Keywords: PG201; Non-inferiority; 100mm pain VAS
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — herbal extract PG201; Celecoxib; Drug Contamination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PG201 tablet (Experimental)
  Interventions: Drug: PG201 tablet
- Celecoxib capsule (Active Comparator)
  Interventions: Drug: Celebrex capsule

INTERVENTIONS:
Drug: PG201 tablet — One PG201 tablet and one celecoxib placebo capsule(after breakfast, in 30minutes), One PG201 tablet and one celecoxib placebo capsule(after dinner, in 30minutes)
  Other Names: botanical drug
  Arms: PG201 tablet
Drug: Celebrex capsule — One celecoxib capsule and one PG201 placebo tablet(after breakfast, in 30minutes), one celecoxib placebo capsule and one PG201 placebo tablet(after dinner, in 30minutes)
  Other Names: chemical drug
  Arms: Celecoxib capsule

SUMMARY:
The objective of this study was to to evaluate the efficacy and safety of PG201 in osteoarthritis patients.

This clinical study was designated to be non-inferiority test with level of significance: 95%, α=0.05. Type 2 error (β) was set as 0.2, and the power of the test was set as 80%. Assuming 20% drop-out rate, the number of subjects required for each treatment group was estimated to be 154, while the total number of subjects required for the study 308.

non-inferiority margin: 8mm

DETAILED DESCRIPTION:
Patients in the PG201 group were prescribed two PG201 tablets per day(BID) and one celecoxib placebo capsule each in the morning and evening per day for 8 weeks.

Patients in the celecoxib group were prescribed celecoxib 200 mg (one 200 mg capsule and one celecoxib placebo capsule) and one PG201 placebo tablet each in the morning and evening per day for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥40 and ≤ 80years of age.
2. Patients who meet the American College of Rheumatology clinical plus radiographic classification criteria for idiopathic osteoarthritis of the knee, which are defined as follow:

   a patient who had knee pain and radiographically diagnosed osteophytes and met at least one of the followings.
   * Age> 50 years.
   * Morning stiffness for less than 30 minutes.
   * Crepitus during movement of the weight-bearing knee.
3. Patients with symptomatic primary osteoarthritis of the knee at least in the last 3 months prior to screening.
4. Patients who received Nonsteroidal antiinflammatory drugs (NSAIDs)/Cyclooxygenase-2 inhibitor for the treatment of arthritis of the knee for at least 5 days a week during 4 weeks prior to screening.
5. Patients who had a score of 100mm pain VAS ≤80 mm at screening.
6. Patients who had a score of 100mm pain VAS ≥50 mm at baseline.
7. Patients should be able and willing to provide the written informed consent.

Exclusion Criteria:

1. Patients with a history of surgery or arthroscopy of the study joint within the previous 6 months.
2. Patients with trauma of study joint within the previous 12 months.
3. Patients with symptomatic hip osteoarthritis, other condition that would interfere with study assessments.
4. Patients with any other type of arthritis, active malignancies or any active GI, cardiovascular, renal, hepatic, neurologic, or psychiatric disease.
5. Patients with a known hypersensitivity or intolerance to Nonsteroidal antiinflammatory drugs (NSAIDs), aspirin or Cyclooxygenase-2 inhibitor.
6. Patients with uncontrollable hypertension.
7. Patients with any of creatinine, bilirubin, Alanine aminotransferase or Aspartate aminotransferase > 1.5 times the Upper Lange of normal at screening.
8. Patients with a history of drug or alcohol abuse.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
100mm Pain VAS reduction | Screening, Day1, Day28

SECONDARY OUTCOMES:
Pain VAS total score on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Screening, Day1, Day28
Sub-scale score and total score on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Screening, Day1, Day28
The change in the quality of life score | Day1, Day28
The change in the patient self-assessed & investigator-assessed overall symptom scores | Screening, Day1, Day28
The responder index (RI) | screening, Day1, Day28

CONTACTS AND LOCATIONS:
Overall Officials: Yeong-wook Song, MD, Principal Investigator — Seoul National University Hospital; Wan-Hee Yoo, MD, Principal Investigator — Chonbuk National University Hospital; Sung-Hwan Park, MD, Principal Investigator — The Catholic University of Korea College of Medicine; Han-joo Baek, MD, Principal Investigator — Gachon University of Medicine and Science; Yun Jong Lee, MD, Principal Investigator — Seoul National University Bundang Hospital; Seung Cheol Shim, MD, Principal Investigator — Eulji University; Seong Wook Kang, MD, Principal Investigator — Chungnam National University School of Medicine; Hyun Ah Kim, MD, Principal Investigator — Hallym University Medical Center; Jung Soo Song, MD, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine; Chang Hee Suh, MD, Principal Investigator — Ajou University School of Medicine; Sung Jae Choi, MD, Principal Investigator — Korea University; Bo Young Yoon, MD, Principal Investigator — Inje University Ilsan Paik Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea